CLINICAL TRIAL: NCT02849054
Title: Optimisation of Neonatal Ventilation: Congenital Diaphragmatic Hernia - Determining the Appropriate Level of Volume Guarantee
Brief Title: CDH - Optimisation of Neonatal Ventilation
Acronym: CDH-ONV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KCH16-080
Record Dates: First submitted 2016-07-18; First posted 2016-07-29 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 4, 5, 6ml/kg targetted tidal volume (Experimental): Randomised to receive TTV at 4ml/kg, 5ml/kg, 6ml/kg. Measurement of PTPdi
  Interventions: Device: Measurement of PTPdi; Device: TTV at 4ml/kg; Device: TTV at 5ml/kg; Device: TTV at 6ml/kg
- 4, 6, 5ml/kg targetted tidal volume (Experimental): Randomised to receive TTV at 4ml/kg, 6ml/kg, 5ml/kg. Measurement of PTPdi
  Interventions: Device: Measurement of PTPdi; Device: TTV at 4ml/kg; Device: TTV at 5ml/kg; Device: TTV at 6ml/kg
- 5, 4, 6ml/kg targetted tidal volume (Experimental): Randomised to receive TTV at 5ml/kg, 4ml/kg, 6ml/kg. Measurement of PTPdi
  Interventions: Device: Measurement of PTPdi; Device: TTV at 4ml/kg; Device: TTV at 5ml/kg; Device: TTV at 6ml/kg
- 5, 6, 4ml/kg targetted tidal volume (Experimental): Randomised to receive TTV at 5ml/kg, 6ml/kg,4ml/kg. Measurement of PTPdi
  Interventions: Device: Measurement of PTPdi; Device: TTV at 4ml/kg; Device: TTV at 5ml/kg; Device: TTV at 6ml/kg
- 6, 5, 4ml/kg targetted tidal volume (Experimental): Randomised to receive TTV at 6ml/kg, 5ml/kg, 4ml/kg. Measurement of PTPdi
  Interventions: Device: Measurement of PTPdi; Device: TTV at 4ml/kg; Device: TTV at 5ml/kg; Device: TTV at 6ml/kg
- 6, 4, 5ml/kg targetted tidal volume (Experimental): Randomised to receive TTV at 6ml/kg, 4ml/kg, 5ml/kg. Measurement of PTPdi
  Interventions: Device: Measurement of PTPdi; Device: TTV at 4ml/kg; Device: TTV at 5ml/kg; Device: TTV at 6ml/kg

INTERVENTIONS:
Device: Measurement of PTPdi — Insertion of pressure transducer catheter to measure gastic and oesophadgeal pressures for calculation of PTPdi
Device: TTV at 4ml/kg — Provision of targetted tidal volume of 4ml/kg
Device: TTV at 5ml/kg — Provision of targetted tidal volume of 5ml/kg
Device: TTV at 6ml/kg — Provision of targetted tidal volume of 6ml/kg

SUMMARY:
To determine the appropriate volume (size) of ventilator breath during volume-targetted ventilation for infants born with congenital diaphragmatic hernia.

ELIGIBILITY:
Inclusion Criteria:

* Congenital diaphragmatic hernia - post-operative Mechanically ventilated Born at >34/40

Exclusion Criteria:

* neuromuscular blockade contraindications to NG/OG tube insertion

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pressure Time Product of the diaphragm (PTPdi) at different levels of targetted tidal volume | 3 hours
  PTPdi will be measured at each level of tidal volume. The outcome measure is the change in PTPdi.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, MD, MBBS, Principal Investigator — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided